CLINICAL TRIAL: NCT04503252
Title: Probability of Target Attainment With Standard Intermittent Bolus Administration of Cefazolin in Patients With Complicated Infections Caused by Staphylococcus Aureus: A Prospective Single-center Cohort Study
Brief Title: Probability of Target Attainment With Standard Intermittent Bolus Administration of Cefazolin in Patients With Complicated Infections Caused by Staphylococcus Aureus
Acronym: TARGET II
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: propatient foundation Basel (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-02229; me20Osthoff2
Record Dates: First submitted 2020-07-29; First posted 2020-08-07 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Staphylococcus Aureus Infection
Keywords: Bloodstream infection (BSI); Minimum inhibitory concentration (MIC); Methicillin-susceptible S. aureus (MSSA); Staphylococcus aureus (S. aureus); β-lactam antibiotics; flucloxacillin; cefazolin; pharmacological target attainment; Torque Teno virus (TTV); Therapeutic drug monitoring (TDM); antibiotic sweat concentrations; Complicated S. aureus infection (CSAI)
MeSH Terms: conditions — Staphylococcal Infections; Sepsis | interventions — Blood Specimen Collection; Sweating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All bacterial isolates from the patients will be stored in the biobank of the microbiology department of the University Hospital Basel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study population: patients with CSAI caused by MSSA: Inpatients with CSAI caused by MSSA treated or intended to receive cefazolin within the next 24-48 hours (at least 10 (maximum of 20) critically-ill patients, at least 10 (maximum of 20) patients with an estimated glomerular filtration rate of <60ml/min, at least 10 patients with BSI).
  Interventions: Other: Blood samples for the measurement of the concentration of cefazolin; Other: S. aureus culture isolate; Other: structured telephone interview
- Sub-study: Torque Teno virus (TTV) viremia: TTV viral load may indicate the immunological status of the host. The TTV sub-study is to to describe the viral kinetics of TTV in CSAI patients.
  Interventions: Other: Blood samples for the measurement of the concentration of cefazolin; Other: S. aureus culture isolate; Other: structured telephone interview; Other: Sub-study quantitative measurement of Torque Teno virus
- Sub-study: cefazolin concentrations in sweat: Out of the study population (patients with CSAI) a total of 15 CSAI patients will be included for the substudy investigating cefazolin concentrations in sweat as a non-invasive therapeutic drug monitoring.
  Interventions: Other: Blood samples for the measurement of the concentration of cefazolin; Other: S. aureus culture isolate; Other: structured telephone interview; Other: Sub-study investigating cefazolin concentrations in sweat

INTERVENTIONS:
Other: Blood samples for the measurement of the concentration of cefazolin — Blood samples for the measurement of the concentration of cefazolin will be collected on the 1st (mid-dose and trough sample), 3rd (mid-dose and trough sample),7th and 14th day (for both only trough sample) of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (usually within 4 weeks after inclusion; only in patients on outpatient continuous parenteral antibiotic treatment).
Other: S. aureus culture isolate — The S. aureus culture isolate will be subjected to exact cefazolin MIC determination and to measurement of the level of cefazolin tolerance.
Other: structured telephone interview — Structured telephone interview for Patient follow- up after 30 days
Other: Sub-study quantitative measurement of Torque Teno virus — An additional EDTA sample will be drawn for quantitative polymerase chain reaction (PCR) of TTV DNA and analyses of cytokines and other parameters of the activation state of the immune system.
  Groups: Sub-study: Torque Teno virus (TTV) viremia
Other: Sub-study investigating cefazolin concentrations in sweat — For each visit of included patients, a sweat sample will be collected via a CE certified Macroduct Sweat Collector. Eccrine sweat glands of the lower forearms are stimulated by pilocarpine (a parasympathomimetic) as well as a local current for 5min. Sweat is subsequently collected by capillary containers during 30min and transferred to small tubes on dry ice. Sweat sample analysis is conducted using mass spectrometry.
  Groups: Sub-study: cefazolin concentrations in sweat

SUMMARY:
Given the paucity of pharmacological data on cefazolin treatment of Methicillin-susceptible S. aureus (MSSA) complicated S. aureus infection (CSAI), the primary purpose of this study is to investigate the probability of pharmacological target attainment (in the blood and infected tissue) with standard intermittent bolus administration of cefazolin in patients with CSAI caused by MSSA by determining plasma concentrations of cefazolin and exact Minimum inhibitory concentration (MICs) of the causative MSSA strains in patients with various disease severities (e.g. critically ill vs. noncritically ill patients).

* Sub-study quantitative measurement of Torque Teno virus (TTV): The primary purpose of this sub-study is to describe the viral kinetics of TTV in CSAI patients and to explore the association of TTV viremia with clinical outcomes and molecular markers of activation of the immune system.
* Sub-study investigating antibiotic concentrations in sweat as a non-invasive therapeutic drug monitoring

ELIGIBILITY:
Inclusion Criteria:

* CSAI caused by MSSA. CSAI is defined as MSSA BSI with a positive follow-up blood culture result for MSSA or the presence of a site of infection remote from the primary focus caused by hematogenous seeding (e.g. endocarditis, vertebral osteomyelitis) or extension of the infection beyond the primary focus (e.g. septic thrombophlebitis or abscess); or deep-seated infections caused by MSSA (e.g. osteoarticular infections, deepseated abscesses).
* Current or intended treatment with cefazolin

Exclusion Criteria:

* Previous enrolment into the current study within 30 days
* Hemodialysis (patients on hemofiltration are eligible)
* Patients who are very likely to stop treatment with cefazolin in the next 48 hours as per treating physician (because of treatment failure, switch to oral medication, palliative care, allergy etc.) or who are very likely to be discharged in the next 48 hours as per treating physician.
* Outpatients
* Women who are pregnant (special pharmacokinetic)
* Polymicrobial infection except concomitant isolation of a likely contaminant (e.g. Staphylococcus epidermidis or Propionibacterium acnes) or an anaerobic pathogen. If an additional pathogen is identified after inclusion of the patient into the study, the patient will remain in the study.
* Not-complicated S. aureus infections: non-bacteremic skin- and soft tissue or small Joint infections without deep-seated abscesses (as these patients will be quickly switched to oral antibiotics)
* CSAI caused by methicillin-resistant S. aureus (MRSA)

Additional exclusion criteria for the sub-study investigating cefazolin concentrations in sweat:

* Allergic to pilocarpine
* Continuous oxygen therapy without the possibility to interrupt oxygen administration for 10min
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with CSAI fulfilling the inclusion criteria and admitted at the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Trough concentration of cefazolin in plasma samples | 1st (mid-dose and trough sample), 3rd (mid-dose and trough sample),7th and 14th day (for both only trough sample) of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  Trough concentration of cefazolin measured in plasma samples
Total plasma concentrations of cefazolin in plasma samples | 1st (mid-dose and trough sample), 3rd (mid-dose and trough sample) of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  Total plasma concentrations of cefazolin in plasma samples
Free drug concentrations of cefazolin in plasma samples | 1st (mid-dose and trough sample), 3rd (mid-dose and trough sample) of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  Free drug concentrations of cefazolin in plasma samples
Trough concentration of cefazolin in sweat samples | 1st, 3rd,7th and 14th day of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  Trough concentration of cefazolin measured in sweat samples
Total sweat concentrations of cefazolin | 1st, 3rd,7th and 14th day of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  Total sweat concentrations of cefazolin
Free drug concentrations of cefazolin in sweat samples | 1st, 3rd,7th and 14th day of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  Free drug concentrations of cefazolin in sweat samples
Target attainment (100%fT>MIC) | 1st, 3rd,7th and 14th day of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  Antibiotic susceptibility of the isolated pathogens determined by the use of an Minimum inhibitory concentration (MIC) test strip. Target attainment (100%fT>MIC) will be calculated for each patient and for each day the patient was sampled. Target attainment is defined as a measured free trough plasma concentration of cefazolin above the measured exact MICs of the causative pathogens at all points of time sampled.

SECONDARY OUTCOMES:
Pharmacological target attainment (100%fT>MIC) in infected tissue | 1st, 3rd,7th and 14th day of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  For the analysis of pharmacological target attainment (100%fT>MIC) in infected tissue (only patients with a suggestive focus or metastatic complication of BSI will be included for this analysis) free trough concentration of cefazolin will be measured in plasma samples.
Attainment of an accepted threshold for toxicity (100%fT>10xMIC) in blood | 1st, 3rd,7th and 14th day of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  For the analysis of attainment of an accepted threshold for toxicity (100%fT>10xMIC) in blood, trough free concentration of cefazolin will be measured in plasma samples. Attainment of the threshold for toxicity is defined as measured free trough plasma concentration of cefazolin above at least 10x the measured exact MIC or above the clinical breakpoint MIC of the causative pathogen as published by the European Committee on Antimicrobial Susceptibility Testing at one time point or more. Cefazolin concentrations in sweat will be compared between patients with attained toxicity and non-attained thresholds in plasma.
Level of cefazolin tolerance of the isolated pathogen | 1st, 3rd,7th and 14th day of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  The level of cefazolin tolerance of the isolated pathogen will be determined by the tolerance disc test as well as through time-kill curves. The level of tolerance determines the required antibiotic concentration to achieve bactericidal killing.
TTV substudy: quantification of DNA | 1st, 3rd,7th and 14th day of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  For the TTV substudy DNA will be extracted from ethylenediaminetetraacetic acid (EDTA) blood and quantified
TTV substudy: quantification of cytokines | 1st, 3rd,7th and 14th day of cefazolin treatment (+/-1-5 day) and if applicable in weekly intervals during outpatient parenteral antibiotic treatment (within 4 weeks)
  Cytokines as a markers of the activation status of the immune system will be quantified by using commercially available ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osthoff, PD Dr. med., Principal Investigator — University Hospital Basel, Division of Internal Medicine
Locations (1):
- University Hospital Basel, Division of Internal Medicine, Basel, Switzerland